CLINICAL TRIAL: NCT00000343
Title: Brain Changes in Stimulant Dependent Subjects
Brief Title: Brain Changes in Stimulant Dependent Subjects - 8
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-3-0010-8; Y01-3-0010-8
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 1996-04

CONDITIONS: Substance-Related Disorders
Keywords: stimulant dependence
MeSH Terms: conditions — Substance-Related Disorders | interventions — Counseling

INTERVENTIONS:
Behavioral: counseling

SUMMARY:
The purpose of this study is to identify the neurophysiologic indicators of cocaine or methamphetamine use and withdrawal, to examine the relationship between subjects' reports of depression, craving, and stimulant use, and neurophysiologic measures, and to identify neurophysiologic measures which can be used to identify new treatments for stimulant dependence.

DETAILED DESCRIPTION:
By Incorporating QEEG into clinical trails, the plan is to develop physiologic markers of treatment efficacy, and to aid in the identification of effective treatments.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Meet DSM-IV criteria for cocaine dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nursing women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90
Dates: Start 1996-04

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States